CLINICAL TRIAL: NCT06714357
Title: Randomized Phase 2 Study of Valproic Acid Combined With Rechallenge Anti-EGFR Based Regimen Regimens in Pretreated Patients With RAS/BRAF Wild-type Metastatic Colorectal Cancer - VICTORIA Trial
Brief Title: ValproIc Acid to Potentiate Anti-EGFR Treatment Efficacy and Prevent/Revert Resistance in Colorectal Cancer
Acronym: VICTORIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICTORIA; 2024-514420-16-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metastatic colorectal cancer; RAS/BRAF wt; Liquid biopsy; Valproic Acid; anti-EGFR treatment; epigenetic reprogramming
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Panitumumab; Valproic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STUDY PART 1 - ARM A - control arm (Active Comparator): Patients will continue to receive standard rechallenge with irinotecan and panitumumab until treatment failure, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria.
  Interventions: Drug: irinotecan; Drug: panitumumab
- STUDY PART 1 - ARM B - experimental arm (Experimental): Patients will continue to receive standard rechallenge with irinotecan and panitumumab in combination with VPA until treatment failure, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria.
  Interventions: Drug: irinotecan; Drug: panitumumab; Drug: Valproic Acid (VPA)

INTERVENTIONS:
Drug: irinotecan — Administered at the dosage of 180 mg/m2 over 60 minutes
Drug: panitumumab — Administered as 60 minutes, or 90 minutes for doses over 1000 mg, intravenous infusion at the dosage of 6 mg/kg
Drug: Valproic Acid (VPA) — VPA will be administered in each patient with a titration strategy to improve the compliance for the treatment, looking for a target serum level between 50 and 100 μg/mL that represents the recommended values for the treatment of epilepsy and also a useful concentration to produce the desired synergistic effect with chemotherapy based on preclinical studies.
  Administrated at the dosage of 500 mg/three times a day (after 7 days of gradual dose escalation).
  Arms: STUDY PART 1 - ARM B - experimental arm

SUMMARY:
The investigators hypothesize that the epigenetic agent valproic acid improve the activity of anti-EGFR agents, prevent and revert the emergence of EGFR resistance, in a rechallenge setting.

Correlative mechanistic studies on tissue and blood samples, liquid biopsies, could identify potential biomarkers of efficacy and help understanding the evolutionary dynamics of tumors in response to therapy thus optimizing the treatment approach with a personalized anti- EGFR treatment strategy.

DETAILED DESCRIPTION:
This study is a multicentric open label academic randomized phase-2 study. The study population will include patients with advanced or metastatic colorectal cancer, RAS/BRAF wt mCRC, eligible for a rechallenge setting (third or later line), with RAS/BRAF wt ctDNA status at study entry. A total of 130 patients (65/arm) will be required.

The VICTORIA - Study Part 1 is a phase 2, open label, randozimed study. Before starting study Part 1 treatment, at the time of enrollment, patients will be randomized electronically 1:1 to one of the two arms: ARM A (standard treatment: irinotecan + panitimumab) and ARM B (VPA + irinotecan + panitumumab) Each cycle will be administered every two weeks for both arms. Patients will continue to receive study treatment until treatment failure as previous defined, unacceptable toxicity, physician's decision, patient's refusal, or any other discontinuation criteria.

All subjects who finish treatment, whichever the reason, will enter in the follow-up. All patients will be followed until death and data on subsequent treatment will be collected.

VPA will be administered per os daily with a titration strategy (table 2 of the protocol) to improve the compliance for the treatment, with a target serum level between 50 and 100 μg/mL that represents the recommended values for epilepsy and also a useful concentration to produce the desired synergistic effect with chemotherapy based on preclinical studies (0.5- 1mM).

An initial safety run-in phase involves a safety evaluation after the first 6 patients are randomly assigned to Arm B. Enrollment will be paused after the first 6 patients randomly assigned to Arm B complete 2 cycles of treatment. The enrollment will be interrupted if the treatment combination will be judged not feasible and major safety concerns will arise. A safety review will be conducted, and recommendations will be made by the Steering Committee. The study will continue if there are 2 or fewer adverse events (AEs) of grade 3 or higher deemed related to the addition of valproic acid to the panitumumab + irinotecan.

All measurable and non-measurable lesions must be documented at screening (within 28 days prior to randomization) and re-assessed at each subsequent tumor evaluation (every 8 weeks). Tumor assessment by CT scan (chest, abdomen and pelvis) or MRI (abdomen and pelvis); CEA, CA 19.9; and any other tests resulted positive during baseline staging, will be performed at week 8 and every 8 weeks during treatment until treatment failure in both arms. Patients discontinuing study treatment without progressive disease, will undergo tumor assessments every 8 weeks until progressive disease or study withdrawal.

Toxicities will be evaluated at each clinical visit throughout the study treatment and up to 4 weeks after last cycle of treatment accordingly to the Common Terminology Criteria for Adverse Events (AEs) of the National Cancer Institute (CTCAE-NCI) version 5.0.

Quality of Life will be assessed by the EORTC QLQ-C30 v.3.0 and QLQ-CR29 questionnaire that will be completed by patients at baseline (prior to treatment, once eligibility is confirmed) and every 8 weeks until disease progression, treatment failure or death. At the same time points will be administered selected items of PRO (Patients Reported Outcome) -CTCAE questionnaire.

Blood samples will be collected at baseline, during treatment, and at progression. Biomarkers will be correlated with clinical response, patient outcome and toxicity. In addition, biomarkers will be evaluated on tumor tissues from primary tumors or metastases at baseline, when available.

To detect a difference between the two groups of 20%; considering 5% of drop out, 61 patients in each arm will be required to achieve 80% power.

A null hypothesis of 0.50 is based on the assumption that the median PFS for RAS wt patients rechallenged with anti-EGFR is approximately 16 weeks. An alternative hypothesis of 0.70 represents a potential target of interest for further studies in this setting with the experimental treatment.

The test statistic used will be the one-sided stratified (for the stratification factors) Fisher's Exact Test. The significance level of the test is targeted at 0.10. The date of end of study will be the date of the last visit of the last patient.

Randomization will be performed with a stratified procedure that will account for tumor sidedness (left vs right), number of metastatic sites (1 vs ≥ 2), previous lines of treatment (2 vs ≥ 3 lines).

The VICTORIA - Study Part 2 is a phase 2, single arm study, designed according to the Fleming single-stage design.

In patients in ARM A, at time of disease progression, a second study will explore if the addition of VPA to irinotecan and panitumumab might revert the occurrence of resistance.

According to the Fleming single-stage design, under the null hypothesis of 0.05, based on the assumption that treatment with standard rechallenge treatment beyond progression usually leads to an extremely low PFS, and under the alternative hypothesis of a PFS rate at 8 weeks of 0.20 with the experimental treatment (a potential target of interest for further studies), considering one-sided alpha and beta errors of 0.05 and 0.20 (80.32) respectively, a total of 27 patients will be required.

A null hypothesis of 0.05 is based on the assumption that treatment beyond PD usually leads to an extremely low PFS. An alternative hypothesis of 0.20 represents a potential target of interest for further studies in this setting with the experimental treatment.

Null hypothesis will be rejected if at least 4 patients will be free of progression at 8 weeks with the experimental treatment.

ELIGIBILITY:
Inclusion Criteria (Study Part 1):

1. Written informed consent to study procedures and to correlative studies.
2. Either sex aged ≥ 18.
3. Histologically proven of colorectal adenocarcinoma.
4. Diagnosis of metastatic disease.
5. RAS/BRAF wild-type status at initial diagnosis assessed at local centers according with a validated method defined by EMA and known MMR/MSI status
6. RAS (NRAS and KRAS exon 2,3 and 4) and BRAF wild-type in liquid biopsy at study entry (according to central testing).
7. Patient candidate to anti-EGFR rechallenge therapy with panitumumab and irinotecan as clinical practice; Efficacy of anti-EGFR drug in any line of treatment with a major response achieved (i.e. complete or partial response according to RECIST criteria v1.1) or stable disease ≥ 6 months and received a subsequent line of therapy upon progression.

   a. Note. Patients must have received at least 2 lines of treatment. Previous treatment with regorafenib, trifluridine/tipiracile, trifluridine/tipiracile + bevacizumab or fruquintinib is allowed. Previous rechallenge with anti-EGFR MoAb is NOT allowed. Adjuvant treatment will be considered as one line of therapy in case of progression within 6 months from the last dose of treatment.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 at study entry.
9. Imaging-documented measurable disease, according to RECIST 1.1 criteria.
10. Estimated life expectancy of more than 12 weeks
11. Adequate bone marrow hematological function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L and platelet count ≥ 100 x 109/L and hemoglobin ≥ 9 g/dL.
12. Adequate liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 2 (in case of biliary stent) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 5 X ULN.
13. Adequate renal function: serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min in males and ≥50 mL/min in females (calculated according to Cockroft-Gault formula).
14. Electrolytes (i.e. magnesium, calcium, sodium and potassium) within laboratory normal range.

Exclusion Criteria (Study Part 1):

1. Prior malignancy within five years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
2. Any contraindication to panitumumab or irinotecan.
3. Not received immunotherapy if dMMR or MSI-H.
4. Patients who have had prior treatment with an HDAC inhibitor and patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid.
5. Major surgical intervention within 4 weeks prior to enrollment.
6. Pregnancy and breast-feeding.
7. Any brain metastasis.
8. Patients with long QT-syndrome or QTc interval duration > 480 msec or concomitant medication with drugs prolonging QTc .
9. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol, or would interfere with the results of the study.
10. History of poor co-operation, non-compliance with medical treatment, unreliability or any condition that may impair the patient's understanding of the Informed consent form.
11. Participation in any interventional drug or medical device study within 30 days prior to treatment start.
12. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.
13. History of interstitial pneumonitis or pulmonary fibrosis.
14. History of corneal perforation or ulceration keratitis.
15. Hypersensitivity to valproic acid or any of listed excipients.
16. Acute hepatitis or chronic hepatitis.
17. Personal or familial anamnesis of severe hepatopathy.
18. History of Hepatic porphyria
19. Known coagulation disorders.
20. Known Polymerase-gamma (POLG) mitochondrial mutation (e.g. Alpers-Huttenlocher Syndrome).
21. Known urea cycle disorders.

    * Inclusion Criteria (Study Part 2):

1. Have provided written informed consent to study procedures and to correlative studies.

2. Enrolled in VICTORIA - Study Part 1 and randomized to ARM A (control arm) 3. Progressed to treatment within ARM A (control arm). 4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 at study entry.

5. Imaging-documented measurable disease, according to RECIST 1.1 criteria. 6. Estimated life expectancy of more than 12 weeks. 7. Adequate bone marrow hematological function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L and platelet count ≥ 100 x 109/L and hemoglobin ≥ 9 g/dL. 8. Adequate liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 2 (in case of biliary stent) and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 5 X ULN. 9. Adequate renal function: serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min in males and ≥50 mL/min in females (calculated according to Cockroft-Gault formula). 10. Electrolytes (i.e. magnesium, calcium, sodium and potassium) within laboratory normal range.

-Exclusion Criteria (Study Part 2):

1. Did not receive a subsequent line of therapy upon progression to ARM A.
2. Any brain metastasis.
3. Pregnancy and breast-feeding.
4. Serious Adverse events with panitumumab or irinotecan, leading to treatment interruption and discontinuation.
5. Patients with long QT-syndrome or QTc interval duration > 480 msec or concomitant medication with drugs prolonging QTc
6. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study, or which would jeopardize compliance with the protocol, or would interfere with the results of the study.
7. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Study Part 1 - Progression Free Survival rate at 16 weeks in the two arms. | up to 16 weeks from randomization
  Progression Free Survival rate at 16 weeks (PFS rate at 16-weeks) is defined as the rate of assessable patients alive and not progressed after 16 weeks from initiation of VICTORIA - Study Part 1 (i.e randomization) to the first documentation of objective disease progression by RECIST 1.1 criteria, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Study Part 1: Progression free survival (PFS) | up to 1 year last patients randomized
  Progression free survival (PFS) calculated as the time from randomization until the date of death from any cause until the date of the first observation of disease progression or death due to any cause, whichever occurs first. PFS will be censored at the time of the last available tumor assessment documenting absence of progressive disease for patients alive at the time of analysis.
Study Part 1 - Overall survival (OS) | up to 1 year last patients randomized
  Overall survival (OS) calculated as the time from randomization until the date of death from any cause. OS will be censored at the last date the patient was known to be alive for patients alive at the time of analysis.
Study Part 1: Objective Tumor Response Rate (ORR) | up to 1 year last patients randomized
  Objective Tumor Response Rate (ORR) assessed according to RECIST criteria 1.1, as the proportion of patients achieving complete or partial response relative to total enrolled patients.
Study Part 1: Disease Control Rate (DCR) | up to 1 year last patients randomized
  Disease Control Rate (DCR) defined as the proportion of patients with complete/partial response and stable disease as their best response.
Study Part 1: Overall Toxicity rate | up to 1 year last patients randomized
  Overall Toxicity rate defined as adverse events graded according NCI CTCAE v 5.0. as the proportion of patients experiencing any grade AE accordingly to the NCI Common Terminology Criteria of Adverse Events (NCI CTC-AE) Version 5, relative to the total of patients receiving at least one cycle of treatment.AE will be listed individually by the patient and summarized overall (severity grades 1-4) and for grade ≥3 by treatment received.
Study Part 1 - Quality of life (QoL) | up the date of first documented progression (assessed up to 1 year)
  Quality of life (QoL) investigated through the EORTC QOL-C30 questionnaires at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks until disease progression, treatment failure or death.
Study Part 1 - Quality of life (QoL) | up the date of first documented progression (assessed up to 1 year)
  Quality of life (QoL) investigated through the CR29 questionnaires at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks until disease progression, treatment failure or death.
Study Part 1 - Quality of life (QoL) | up the date of first documented progression (assessed up to 1 year)
  Quality of life (QoL) investigated through the PRO-CTCAE questionnaire at baseline (prior to treatment start, once eligibility is confirmed) and every 8 weeks until disease progression, treatment failure or death.

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - AORN Sant'Anna e San Sebastiano, Caserta, CE
  - Università degli studi della Campania Luigi Vanvitelli, Napoli, Italia
  - AORN San Giuseppe Moscati Avellino, Avellino, Italy
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, Italy
  - Pia Fondazione Di Culto E Religione Card G Panico, Tricase, Lecce
  - Ospedale Civile San Giovanni di Dio, Frattamaggiore, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Napoli
  - Presidio Ospedaliero "Santa Maria delle Grazie", Pozzuoli, PZ